CLINICAL TRIAL: NCT01330173
Title: A Phase 1b Study of GDC-0449 Following Autologous Transplantation in Patients With High Risk First Remission or Relapsed Multiple Myeloma
Brief Title: Vismodegib After Stem Cell Transplant in Treating Patients With High-Risk First Remission or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02914; NCI-2012-02914 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00040967; JHOC-J1067; NA_00040967 / J1067; CDR0000691708; J1067 (Other: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital); 8414 (Other: CTEP); U01CA070095 (NIH); UM1CA186691 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-09

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — HhAntag691

ARMS (1):
- Treatment (vismodegib) (Experimental): Patients receive vismodegib PO QD on days 1-28. Treatment repeats every 28 days for up to 11 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Vismodegib; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies how well vismodegib after stem cell transplant works in treating patients with high-risk first remission or relapsed multiple myeloma. Vismodegib may slow the growth of cancer cells. Giving vismodegib after autologous stem cell transplant may kill more multiple myeloma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if GDC-0449 (vismodegib) is able to reduce myeloma cancer stem cells (CSC) when given to patients with multiple myeloma (MM) following autologous stem cell transplantation.

SECONDARY OBJECTIVES:

I. To determine whether GDC-0449 is inhibiting the hedgehog (Hh) pathway in patients with MM following autologous transplantation by measuring downstream targets of Hh using quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) on plasma cells and MM CSC obtained from blood and bone marrow of patients undergoing treatment.

II. To determine whether changes in MM CSC as measured by clonogenic assays on bone marrow are seen in response to GDC-0449 and whether these changes predict recurrence.

III. To determine whether changes in MM CSC can be measured with similar or better accuracy using peripheral blood flow cytometry as compared to bone marrow clonogenic assays.

IV. To determine the safety and toxicity profile for treatment with GDC-0449 following autologous transplantation in patients with high risk or relapsed MM.

V. To characterize the pharmacokinetics (PK) of GDC-0449 (total and unbound) at steady-state and correlate this with pharmacodynamic (PD) endpoints.

VI. To determine the one year progression free survival for patients given GDC-0449 following autologous transplantation.

OUTLINE:

Patients receive vismodegib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 11 courses in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed multiple myeloma meeting criteria with symptomatic disease requiring treatment; patients considered to have high risk disease (defined as chromosome 13 deletion by cytogenetics; t(4;14), t(14;16) or 17p deletion by fluorescence in situ hybridization [FISH], B2-M > 5.5 g/dL, immunoglobulin A [IgA] phenotype) in first remission (>= partial remission [PR]) or patients with relapsed myeloma responding to salvage therapy (>= PR) based on the International Uniform Response Criteria are eligible
* Patients must have measurable disease utilizing serum or urine protein electrophoresis or serum kappa / lambda light chain assay
* Patients must be planning to proceed to single autologous transplantation according to institutional standards and must receive this transplantation prior to implementation of GDC-0449
* Concomitant bisphosphonate use is allowed as clinically indicated
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to GDC-0449 treatment, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient understands of GDC-0449 cause serious or life-threatening birth defects
  * Women of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had a tubal ligation
  * Women are considered not to be of childbearing potential for the following reasons:

    * The patient has undergone hysterectomy and/or bilateral oophorectomy
    * The patient is post-menopausal defined by amenorrhea for at least 1 year in a women
* Human immunodeficiency virus (HIV)-positive patients without a prior acquired immune deficiency syndrome (AIDS)-defining illness and a CD4 count 400/millimeter^3 and either do not require anti-HIV therapy or are taking anti-HIV therapy that would not interfere with GDC-0449 (e.g. not taking zidovudine, protease inhibitors or non-nucleoside reverse transcriptase inhibitors) are eligible
* Ability to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in MM CSC counts | Baseline to 6 months
  Estimated using a simple linear regression model. The proportion of patients with negative slope estimates, indicating decline in MM CSC counts over study evaluations will be estimated.

SECONDARY OUTCOMES:
Pharmacokinetics of vismodegib | Days 1 and 15
Pharmacodynamics of vismodegib | Up to 4 weeks after completion of study treatment
Time to progression | From treatment initiation to the date of progression, assessed up to 4 weeks after completion of study treatment
  Estimated based on Kaplan-Meier and compared using the nonparametric, log-rank test, with proportional hazards regression used to model the effect of other correlations on the outcome of progression free survival (PFS). Median PFS will reported along with hazard ratios and corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Huff, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital
Locations (2):
- United States (2):
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland